CLINICAL TRIAL: NCT03238287
Title: Evaluation of Effectiveness of Cardiopulmonary Resuscitation With Manual and Mechanical Chest Compression Systems During In-hospital (at the Emergency Department) Witnessed Cardiac Arrests Using Cerebral Oximetry
Brief Title: Manual and Mechanical Chest Compression During In-hospital Witnessed Cardiac Arrests Using Cerebral Oximetry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Collaborators: Scientific Research Projects Commission of ESOGU (Unknown)
Responsible Party: Principal Investigator, Filiz Baloglu Kaya, Ass.Prof., Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 3939444; 2016-1385 (Other Grant/Funding Number: Scientific Research Projects Commission of ESOGU)
Record Dates: First submitted 2017-07-25; First posted 2017-08-03 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Cardiopulmonary Resuscitation
Keywords: Emergency; Mechanical chest compression; Cerebral oximetry
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manuel chest compression (Active Comparator): In the application of advanced cardiac life support, chest compression is done with hands. rSO2 measurements are used to detect the impact of the compression on brain perfusion. The application is performed in accordance with the recommendations on advanced cardiac life support in the current guidelines.
  Interventions: Other: Manuel chest compression
- Mechanical chest compression (Active Comparator): In the application of advanced cardiac life support, chest compression is done with mechanical chest compression device. rSO2 measurements are used to detect the impact of the compression on brain perfusion. The application is performed in accordance with the recommendations on advanced cardiac life support in the current guidelines.
  Interventions: Device: Mechanical chest compression

INTERVENTIONS:
Device: Mechanical chest compression — In the application of advanced cardiac life support, chest compression is done with mechanical chest compression device. rSO2 measurements are used to detect the impact of the compression on brain perfusion. The application is performed in accordance with the recommendations on advanced cardiac life support in the current guidelines.
  Other Names: LUCAS2
  Arms: Mechanical chest compression
Other: Manuel chest compression — In the application of advanced cardiac life support, chest compression is done with hands. rSO2 measurements are used to detect the impact of the compression on brain perfusion. The application is performed in accordance with the recommendations on advanced cardiac life support in the current guidelines
  Arms: Manuel chest compression

SUMMARY:
Post-resuscitation neurological impairment is associated with morbidity and especially with late mortality. Thus, because good neurological outcome is vital for a successful resuscitation, it is essential to have sufficient cerebral tissue perfusion and oxygenation during its application. Near-Infrared Spectroscopy (NIRS) is used to evaluate such conditions. NIRS is a non-invasive technique which provides real-time, continuous information about regional cerebral tissue oxygen saturation levels (regional SO2/rSO2). Research on NIRS has been done in many studies including cardiovascular surgery, neurosurgery and their intensive care processes and its effectiveness has been approved. However, there is limited data on its use in cardiac arrests.

As stated in the current guidelines, sufficient speed and depth of chest compressions, few interruptions of compressions are key to a successful outcome of resuscitation. The studies with the mechanical chest compression devices showed that the earlier it was applied in out-of-hospital cases, the higher the rates of survival until hospitalization. There is not sufficient number of studies on the routine use of mechanical chest compression devices for in-hospital cases. In case the application of manual resuscitation is not convenient (during patient relocation, procedure at the angiography laboratory, and rush hours of emergency services when staff might fall short), alternative methods will be required.

The aim of our study is to compare rSO2 levels measured during resuscitation with manual and mechanical devices in in-hospital (at the emergency department) witnessed cardiac arrest cases and to analyze the impact of both application method and perfusion levels on survival and neurological outcome.

DETAILED DESCRIPTION:
The study will be a single-center, prospective and randomized study. It will be conducted at the Emergency Department of Eskisehir Osmangazi University Education, Application and Research Hospital.

Patients will be allocated to treatment groups by blocked randomization (www.randomizer.org). Advanced cardiac life support algorithm will be initiated as outlined in the current resuscitation guidelines and cardiopulmonary resuscitation (CPR) will be continued either manually or mechanically (with the chest compression system), according to the randomization scheme. Due to the nature of the interventions carried out in the study process, blinding of healthcare providers was not possible.

Before the initiation of the study, the team members participating in the study will receive theoretical and practical training on CPR, mechanical chest compression system utilization and NIRS.

Patients who develop cardiopulmonary arrest during their clinical evaluation in the emergency department will receive CPR, and the chest compression method will be determined by the senior physician according to the randomization scheme.

1. The manual CPR group will receive chest compressions, respiratory support and medical treatment in accordance with the recommendations of current guidelines. If return of spontaneous circulation (ROSC) is achieved, post-resuscitation care will be provided. If ROSC is not achieved, CPR will be terminated in accordance with the recommendations of current guidelines.
2. The patients on the mechanical chest compression group will receive manual chest compressions until the mechanical compression device is installed (about 15-20 seconds). In this time interval, thorax and sternum measurements will be evaluated for suitability for the study, and mechanical compression device will be installed on patients who are deemed suitable. The patients will receive chest compressions, respiratory support and medical treatment in accordance with the recommendations of current guidelines. If ROSC is achieved, post-resuscitation care will be provided. If ROSC is not achieved, CPR will be terminated in accordance with the recommendations of current guidelines.

The presence of ROSC or the decision to terminate CPR will be determined according to the vital signs (arterial blood pressure, heart rate, oxygen saturation with pulse oximeter), end tidal carbon dioxide (ETco2) measurement (with the module device used for the measurement of rSO2) and cardiac assessment with bedside ultrasonography (Vivid e, General Electric Healthcare, China).

As soon as cardiopulmonary arrest is identified, sensors measuring the value of rSO2 will be placed on the patient's head bifrontally (forehead area) in order to measure the cerebral perfusion. During CPR, rSO2 values will be continuously recorded. The placement of the sensors and the measurements will be carried out by a medical staff who received necessary training prior to the study. In order not to affect the clinical decisions made during CPR, the rSO2 device will be placed in a convenient area which is out of the CPR performers' eyesight.

Arterial blood pressure, heart rate, respiratory rate, body temperature, oxygen saturation on pulse oximeter, primary arrest rhythm, any known diseases (if existent) and defibrillation attempts (if existent) will be recorded on the case report form during CPR.

In patients with ROSC, 6-hour and 24-hour survival after CPR, discharge from the hospital with favorable neurologic outcome and the presence of additional pathologies (such as heart failure and neurologic sequelae) will be evaluated. Favorable neurologic outcome was defined as a Cerebral Performance Category score of 1-2. In patients with ROSC, post-resuscitation care will be provided as recommended in the current guidelines.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. In hospital (emergency service) witnessed cardiac arrest.
3. Cardiac arrest caused reasons other than trauma.
4. Length of sternum between 170- 303 mm (devise requirements).
5. Patients' chest width not more than 449 mm (devise requirements).
6. Informed consent of first-degree relatives of patients.

Exclusion Criteria:

1. Younger than 18 years old.
2. Out-of-hospital cardiac arrest.
3. Exposure to trauma.
4. Pregnancy.
5. Length of sternum not between 170- 303 mm (devise requirements).
6. Patients' chest width more than 449 mm (devise requirements).
7. Intracranial mass, large infarct or bleeding in the frontal part of the head (rSO2 monitoring area) which might effect the evaluation.
8. Lack of informed consent of first-degree relatives of patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2019-01-04 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Regional cerebral tissue oxygen saturation level | 20-45 second
  Comparison of regional cerebral tissue oxygen saturation levels between two groups during cardiopulmonary resuscitation

SECONDARY OUTCOMES:
Survival at the 6th hour and 24th hour after resuscitation, | 6th hour and 24th hours
  Survival at the 6th hour and 24th hour after resuscitation and evaluation of neurological outcome (cerebral performance category scale 1-2)
Hospital discharge | 1- 30 days
  Hospital discharge with good neurological outcome (cerebral performance category scale 1-2)
Additional pathology | 1- 30 days
  Evaluation of additional pathology (e.g., renal failure and cardiac failure) after resuscitation during in-hospital observation.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Baloğlu Kaya, Study Chair — Eskisehir Osmangazi University
Locations (1):
- Eskisehir Osmangazi University Medical School, Eskişehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participants data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Data will be available within one year of study completion.
Access Criteria: Data access requests will be reviewed by the principal investigator of the study. Requestors will be required to sign a Data Access Agreement.

REFERENCES:
- [Derived] Baloglu Kaya F, Acar N, Ozakin E, Canakci ME, Kuas C, Bilgin M. Comparison of manual and mechanical chest compression techniques using cerebral oximetry in witnessed cardiac arrests at the emergency department: A prospective, randomized clinical study. Am J Emerg Med. 2021 Mar;41:163-169. doi: 10.1016/j.ajem.2020.06.031. Epub 2020 Jun 28. PMID 33071075